CLINICAL TRIAL: NCT02670538
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Fixed-Dose Clinical Trial Evaluating The Efficacy, Safety And Tolerability Of Cariprazine In Patients With Bipolar I Depression
Brief Title: Study of the Efficacy of a Fixed-dose Regimen of Cariprazine Compared to Placebo for Treatment of the Depressive Episode in Participants With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGH-MD-53; 2016-000756-98 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-02

CONDITIONS: Bipolar Disorder; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cariprazine 3.0 mg (Experimental): Following a 7 to 14 days screening/washout period, cariprazine 1.5 milligrams (mg) capsule, one per day, orally for 2 weeks increased to cariprazine 3.0 mg capsule, one per day orally beginning on Day 15 for 4 weeks.
  Interventions: Drug: Cariprazine
- Cariprazine 1.5 mg (Experimental): Following a 7 to 14 days screening/washout period, cariprazine 1.5 mg capsule, one per day, orally for 6 weeks.
  Interventions: Drug: Cariprazine
- Placebo (Placebo Comparator): Following a 7 to 14 days screening/washout period, matching placebo capsule, one per day, orally for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cariprazine — Cariprazine capsule one per day orally.
  Other Names: Vraylar
  Arms: Cariprazine 1.5 mg; Cariprazine 3.0 mg
Drug: Placebo — Matching placebo capsule one per day orally.
  Arms: Placebo

SUMMARY:
This study is designed to prospectively confirm the efficacy of a fixed-dose regimen of cariprazine 1.5 milligrams (mg)/day or 3 mg/day compared to placebo for treatment of the depressive episode in participants with bipolar I disorder. The safety and tolerability of the fixed-dose regimens will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Currently meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for bipolar I disorder without psychotic features confirmed by the administration of the Mini International Neuropsychiatric Interview (MINI), with a current major depressive episode of at least 4 weeks and not exceeding 12 months in duration
* Currently treated as an outpatient at the time of enrollment
* A verified previous manic or mixed episode. Verification must include one of the following sources:

  * Treatment of mania with an anti-manic agent (eg, lithium or divalproate) or antipsychotic medication with an approved indication for mania
  * Hospital records/Medical records
  * Patient report corroborated by caretaker or previous or current treating clinician
* 17-item Hamilton Depression Rating Scale (HAMD-17) total score ≥ 20
* HAMD-17 item 1 score ≥ 2
* CGI-S score ≥ 4
* Negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test (women of childbearing potential only)
* Normal physical examination, clinical laboratory test results, and electrocardiogram (ECG) results or abnormal findings that are judged not clinically significant by the Principal Investigator (PI)

Exclusion Criteria:

* Young Mania Rating Scale (YMRS) total score > 12
* Four or more episodes of a mood disturbance (depression, mania, hypomania, or mixed state) within the 12 months before Visit 1
* Any current axis 1 psychiatric diagnosis other than bipolar disorder with the exception of specific phobias
* History of meeting DSM-5 criteria for:

  * Dementia, amnesic, or other cognitive disorder
  * Schizophrenia, schizoaffective, or other psychotic disorder
  * Mental retardation
* DSM-5-based diagnosis of borderline or antisocial personality disorder or other axis II disorder of sufficient severity to interfere with participation in this study
* History of meeting DSM-5 criteria for alcohol or substance abuse or dependence (other than nicotine or caffeine) within the 6 months before Visit 1
* Positive result on blood alcohol test or urine drug screen for any prohibited medication. Exception:

  * Patients with a positive cannabinoid on entry may be retested before randomization. If the patient remains positive, the patient is no longer eligible
  * Patients positive for opiates on entry, discussion with Study Physician is required.
* Electroconvulsive therapy in the 3 months before Visit 1
* Previous lack of response to electroconvulsive therapy
* Treatment with a depot antipsychotic drug within 1 treatment cycle before Visit 1
* Treatment with clozapine in a dose of > 50 mg/day in the past 2 years
* Prior participation in any investigational study of RGH-188 or cariprazine within the past 12 months
* Previous treatment with vagus nerve stimulation or transcranial magnetic stimulation within 6 months before Visit 1
* Prior participation with any clinical trials, involving experimental or investigational drugs, within 6 months before Visit 1 or during the study
* Initiation or termination of psychotherapy for depression within the 3 months preceding Visit 1, or plans to initiate, terminate, or change such therapy during the course of the study.
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
* Gastric bypass or any condition that would be expected to affect drug absorption (lap band procedures are acceptable if there is no problem with absorption)
* Known history of cataracts or retinal detachment
* Known human immunodeficiency virus infection
* Employee, or immediate relative of an employee, of the Sponsor, any of its affiliates or partners, or the study center

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 493 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2018-01-18 (Actual); Study Completion 2018-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Willie Earley, Study Director — Allergan
Locations (89):
- United States (42):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Harmonex Neuroscience Research, Inc., Dothan, Alabama
  - NoesisPharma, LLC, Phoenix, Arizona
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - Advanced Research Center, Inc, Anaheim, California
  - Radiant Research, Cerritos, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Excell Research, Inc., Oceanside, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Comprehensive Clinical Research, Washington D.C., District of Columbia
  - CNS Clinical Research Group, Coral Springs, Florida
  - MD Clinical, Hallandale, Florida
  - Innovative Clinical Research, Inc., Lauderhill, Florida
  - Innova Clinical Trials, Inc., Miami, Florida
  - Research Centers of America, LLC, Oakland Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Baber Research Group, Naperville, Illinois
  - J. Gary Booker, MD, APMC, Shreveport, Louisiana
  - Coastal Research Associates, Inc., Weymouth, Massachusetts
  - Millennium Psychiatric Associates, Creve Coeur, Missouri
  - St. Louis Clinical Trials, LLC, St Louis, Missouri
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Pharmaceutical Research Associates, Inc., Marlton, New Jersey
  - Brooklyn Medical Institute, Brooklyn, New York
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - University at Buffalo Erie County Medical Center, Buffalo, New York
  - Manhattan Behavioral Medicine, New York, New York
  - Eastside Comprehensive Medical Center, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Clinical Trials of America, Inc, Hickory, North Carolina
  - University of Cincinnati - Department of Psychiatry and Behavioral Neuroscience, Cincinnati, Ohio
  - Professional Psychiatric Services, Mason, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Tulsa Clinical Research, LLC, Tulsa, Oklahoma
  - Suburban Research Associates, Media, Pennsylvania
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - Houston Endoscopy and Research Center, Houston, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Pacific Institute of Medical Sciences, Bothell, Washington
- Bulgaria (6):
  - Mental Health Centre 'Prof. Dr. Ivan Temkov', EOOD, Burgas
  - MHAT "Dr. Hristo Stambolski", EOOD, Kazanlak
  - UMHAT 'Dr. Georgi Stranski', Dept. of Psychiatry, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - DCC "Mladost M" - Varna, OOD Site 188, Varna
  - DCC "Mladost M" - Varna, OOD Site 194, Varna
- Croatia (6):
  - Neuropsychiatric Hospital Ivan Barbot, Popovača
  - Clinical Hospital Center Rijeka, Rijeka
  - Polyclinic Neuron, Zagreb
  - University Hospital Center Zagreb, Zagreb
  - Clinic for Psychiatry Vrapce, Zagreb
  - Psychiatric Hospital "Sveti Ivan", Zagreb
- Barbara Diaz-Hernandez MD Research, Inc., San Juan, Puerto Rico
- Romania (5):
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila", Bucharest
  - Spitalul de Psihiatrie Titan "Dr. Constantin Gorgos", Bucharest
  - Spitalul de Psihiatrie "Elisabeta Doamna" Galati, Galati
  - Institutul de Psihiatrie Socola Iasi Site 111, Iași
  - Institutul de Psihiatrie Socola Iasi Site 113, Iași
- Serbia (11):
  - Clinic of Psychiatric Diseases "Dr Laza Lazarevic", Belgrade
  - Clinical Center of Serbia, Belgrade
  - Clinical Center Zvezdara, Belgrade
  - General Hospital Euromedic, Belgrade
  - Institute of Mental Health, Belgrade
  - Clinical Center "Dr. Dragisa Misovic", Belgrade
  - Clinical Center Kragujevac Site 154, Kragujevac
  - Clinical Centre Kragujevac Site 158, Kragujevac
  - Clinical Center Nis Site 150, Niš
  - Clinical Center Nis Site 160, Niš
  - Specialized Hospital for Neuropsychiatric Diseases "Sveti Vracevi", Novi Kneževac
- Slovakia (6):
  - Centrum zdravia R.B.K. s.r.o., Bardejov
  - Vavrusova Consulting s.r.o., Bratislava
  - Liptovska nemocnica s poliklinikou Liptovsky Mikulas, Liptovský Mikuláš
  - PsychoLine s.r.o., Rimavská Sobota
  - Nemocnica s poliklinikou sv. Barbory, Roznava a.s., Rožňava
  - Crystal Comfort s.r.o., Vranov nad Topľou
- Ukraine (12):
  - CI of Kyiv Reg.Council Reg.Psychiatric-Narcological Medical Association, Hlevakha
  - Regional Psychoneurological Hospital #3, Dept of Primary Psych Episode, Ivano-Frankivsk
  - Regional Psychoneurological Hospital #3, Ivano-Frankivsk
  - SI Inst.of Neurology, Psychiatry and Narcology of NAMS of Ukraine, Kharkiv
  - CI Kherson Reg. Psychiatric Hospital of Kherson RC, Kherson
  - CI Odesa Regional Psychiatric Hospital # 2, Komintern
  - CI of LRC Lviv Reg. Council Lviv Reg.Clinical Psychoneurological Dispensary, Lviv
  - CI Odesa Regional Medical Center of Mental Health, Odesa
  - CI Cherkasy Regional Psychiatric Hospital of ChRC, Smila
  - Ternopil Reg. Communal Clinical Psychoneurological Hospital Depts of Psychiatry #2, Ternopil
  - Transcarpathian Regional Narcological Dispensary, Uzhhorod
  - CI O.I. Yushchenko Vinnytsia Reg. Psychoneurological Hospital, Vinnytsia

REFERENCES:
- [Derived] McIntyre RS, Llorca PM, Aronin LC, Yu J, Nguyen HB. Effect of Cariprazine on Anhedonia in Patients with Bipolar I Depression: Post Hoc Analysis of Three Randomized Placebo-Controlled Clinical Trials. Adv Ther. 2025 Jan;42(1):246-260. doi: 10.1007/s12325-024-03009-2. Epub 2024 Nov 9. PMID 39520655
- [Derived] Citrome L, Yatham LN, Patel MD, Barabassy A, Hankinson A, Earley WR. Cariprazine and akathisia, restlessness, and extrapyramidal symptoms in patients with bipolar depression. J Affect Disord. 2021 Jun 1;288:191-198. doi: 10.1016/j.jad.2021.03.076. Epub 2021 Mar 31. PMID 33915374
- [Derived] Thase ME, Harrington A, Calabrese J, Montgomery S, Niu X, Patel MD. Evaluation of MADRS severity thresholds in patients with bipolar depression. J Affect Disord. 2021 May 1;286:58-63. doi: 10.1016/j.jad.2021.02.043. Epub 2021 Feb 20. PMID 33677183
- [Derived] Yatham LN, Vieta E, McIntyre RS, Jain R, Patel M, Earley W. Broad Efficacy of Cariprazine on Depressive Symptoms in Bipolar Disorder and the Clinical Implications. Prim Care Companion CNS Disord. 2020 Sep 17;22(5):20m02611. doi: 10.4088/PCC.20m02611. PMID 32942346
- [Derived] Earley WR, Burgess M, Rekeda L, Hankinson A, McIntyre RS, Suppes T, Calabrese JR, Yatham LN. A pooled post hoc analysis evaluating the safety and tolerability of cariprazine in bipolar depression. J Affect Disord. 2020 Feb 15;263:386-395. doi: 10.1016/j.jad.2019.11.098. Epub 2019 Nov 22. PMID 31969269
- [Derived] Earley WR, Burgess MV, Khan B, Rekeda L, Suppes T, Tohen M, Calabrese JR. Efficacy and safety of cariprazine in bipolar I depression: A double-blind, placebo-controlled phase 3 study. Bipolar Disord. 2020 Jun;22(4):372-384. doi: 10.1111/bdi.12852. Epub 2019 Nov 6. PMID 31628698

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Following a 7 to 14 day screening/washout period, matching placebo capsule, one per day, orally for 6 weeks.
- Cariprazine 1.5 mg: Following a 7 to 14 day screening/washout period, cariprazine 1.5 mg capsule, one per day, orally for 6 weeks.
- Cariprazine 3.0 mg: Following a 7 to 14 day screening/washout period, cariprazine 1.5 mg capsule, one per day, orally for 2 weeks increased to cariprazine 3.0 mg capsule, one per day orally beginning on Day 15 for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Started | 167 | 168 | 158
Safety Population : Received Study Drug | 165 | 167 | 158
Intent-to-Treat Population | 163 | 162 | 153
Completed | 135 | 136 | 128
Not Completed | 32 | 32 | 30
Not completed — Withdrawal of Consent | 8 | 6 | 5
Not completed — Lost to Follow-up | 8 | 12 | 7
Not completed — Adverse Event | 5 | 5 | 11
Not completed — Lack of Efficacy | 7 | 1 | 2
Not completed — Protocol Violation | 3 | 4 | 1
Not completed — Noncompliance with Study Drug | 1 | 3 | 2
Not completed — Other Miscellaneous Reasons | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Randomized Population consisted of all participants in the Screened Population who were randomized to a treatment group in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg | Total
Number analyzed (Participants) | 167 | 168 | 158 | 493
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (11.6) | 42.2 (12.0) | 43.9 (11.8) | 43.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 107 | 103 | 309
  Male | 68 | 61 | 55 | 184
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 121 | 121 | 117 | 359
  Black or African American | 46 | 41 | 39 | 126
  Asian | 0 | 3 | 2 | 5
  Multiple Races | 0 | 3 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 22 | 15 | 55
  Not Hispanic or Latino | 149 | 146 | 143 | 438
Montgomery-Åsberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: score on a scale] — MADRS is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants were rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each of the 10 items was scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity for a total possible score of 0 (best) to 60 (worst). Population: Intent-to-Treat (ITT) Population consisted of all participants in Safety Population who had at least 1 postbaseline assessment of MADRS total score.
  score on a scale
    number analyzed (Participants) | 163 | 162 | 153 | 478
    (all) | 31.4 (4.5) | 31.5 (4.3) | 31.5 (4.8) | 31.5 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS)
Description: MADRS is a 10-item, clinician-rated scale that evaluates the participants depressive symptomatology during the past week. Participants were rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each of the 10 items was scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity for a total possible score of 0 (best) to 60 (worst). A negative change from Baseline indicates improvement. Mixed-effects Model for Repeated Measures (MMRM) with fixed factors (treatment group, pooled study center, and visit), baseline (a covariate), and interactions (treatment group by visit, baseline by visit).
Time Frame: Baseline (Week 0) to Week 6
Population: ITT Population consisted of all participants in Safety Population who had at least 1 postbaseline assessment of MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Number analyzed (Participants) | 163 | 162 | 153
score on a scale | -12.4 (0.75) | -14.8 (0.76) | -14.1 (0.78)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 1.5 mg; Test type: Superiority; p = 0.0417, Contrast t-test — Adjusted p-value: adjustment was performed using matched parallel gatekeeping procedure to control the overall type I error rate for multiple comparisons of 2 active doses versus placebo at Week 6; Least Squares (LS) Mean Difference = -2.5, 95% CI 2-sided [-4.6 to -0.4]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 3.0 mg; Test type: Superiority; p = 0.1051, Contrast t-test — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -1.8, 95% CI 2-sided [-3.9 to 0.4]

2. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) Score
Description: CGI-S is a clinician-rated scale that measures the overall severity of a participant's illness in comparison with the severity of other patients the physician has observed. The participant was rated on a scale from 1 to 7, with 1 indicating a "normal state" and 7 indicating "among the most extremely ill patients". A negative change from Baseline indicates improvement. MMRM with fixed factors (treatment group, pooled study center, and visit), baseline (a covariate), and interactions (treatment group by visit, baseline by visit).
Time Frame: Baseline (Week 0) to Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Number analyzed (Participants) | 163 | 162 | 153
score on a scale | -1.2 (0.09) | -1.5 (0.09) | -1.4 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 1.5 mg; Test type: Superiority; p = 0.0417, Contrast t-test — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.3, 95% CI 2-sided [-0.6 to -0.1]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 3.0 mg; Test type: Superiority; p = 0.1370, Contrast t-test — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = -0.2, 95% CI 2-sided [-0.4 to 0.1]

ADVERSE EVENTS:
Time Frame: First dose of study drug up to Day 50
Description: Safety Population, all participants in the Randomized Population who took at least 1 dose of double-blind investigational product, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/167 | 0/158
Serious Adverse Events (participants affected / at risk) | 5/165 | 1/167 | 1/158
Other Adverse Events (participants affected / at risk) | 36/165 | 45/167 | 45/158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=165) | Cariprazine 1.5 mg (N=167) | Cariprazine 3.0 mg (N=158)
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0/97 | 0/107 | 1/103
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Mania (Psychiatric disorders) | 1 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=165) | Cariprazine 1.5 mg (N=167) | Cariprazine 3.0 mg (N=158)
Nausea (Gastrointestinal disorders) | 5 | 13 | 8
Fatigue (General disorders) | 2 | 9 | 5
Akathisia (Nervous system disorders) | 3 | 9 | 15
Headache (Nervous system disorders) | 14 | 14 | 14
Insomnia (Psychiatric disorders) | 7 | 8 | 11
Restlessness (Psychiatric disorders) | 5 | 4 | 11
Agitation (Psychiatric disorders) | 10 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT02670538/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02670538/SAP_001.pdf